CLINICAL TRIAL: NCT02030808
Title: Target-Controlled Infusion of Remifentanil Without Muscle Relaxant Allows Acceptable Surgical Conditions During Thoracotomy
Brief Title: Remifentanil Without Muscle Relaxant for Thoracotomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anesth-Dec13(2)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Elective Open Thoracotomy
Keywords: Thoracic surgery; non-muscle relaxant; target-controlled infusion; remifentanil; surgical conditions
MeSH Terms: interventions — Population Groups; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Muscle Relaxants (MR) group (Placebo Comparator): Cisatracurium will be administered
  Interventions: Drug: Muscle Relaxants (MR) group
- Non- Muscle Relaxants (NMR) group (Active Comparator): No cisatracurium will be administered
  Interventions: Drug: Non- Muscle Relaxants (NMR) group

INTERVENTIONS:
Drug: Muscle Relaxants (MR) group — patients received 0.2 mL/kg cisatracurium® (Nimbex) 0.2%, and a left-sided endobronchial double-lumen tube was placed when the TOF revealed one or two twitches
  Arms: Muscle Relaxants (MR) group
Drug: Non- Muscle Relaxants (NMR) group — No cisatracurium® (Nimbex) will be administered
  Arms: Non- Muscle Relaxants (NMR) group

SUMMARY:
Although the administration of muscle relaxation is essential standard of care for thoracic procedures, it could cause long-reversal times and postoperative residual curarization (PORC) increasing length of post-anesthesia care unit (PACU) stay and hospital costs. Sugammadex offers new perspectives to reduce the incidence of PORC. Unfortunately it is not available in many countries because of its significantly high cost. We hypothesized that the use of target-controlled remifentanil infusion (TCI) with the non-muscle relaxant (NMR) would be associated with comparable surgical conditions and reduced total costs compared with the use of neuromuscular blockers during thoracotomy.

After ethical approval, 66 patients scheduled for elective thoracotomy under sevoflurane anesthesia with TCI remifentanil will be included in this prospective, randomized, single-blind, controlled study.

Patients will be randomly assigned to receive cisatracurium or saline (n = 33 for each group) throughout the procedure. Laryngoscopy and intubating conditions, intraoperative modified thoracic surgery rating scale (Table below), incidence of light anesthesia, and use of vasopressors and anesthetics, clinical recovery, incidence of PORC, PACU and hospital stays, and total costs will be recorded.

DETAILED DESCRIPTION:
Administration of muscle relaxation is essential standard of care in thoracic surgery as it causes an improvement of surgical conditions. The concept of "Fast-track thoracic anesthesia" requires the use of either short or intermediate-acting nondepolarising neuromuscular blocking drugs, to provide a sufficient neuromuscular blockade during surgery and to restore the normal neuromuscular transmission immediately at the end of surgery.1

However, long-reversal times and postoperative residual curarization (PORC) are still a problem in 30%-60% of the anesthetized patients even with the use of new intermediate-acting neuromuscular blockers.2-3 PORC could cause aspiration of the lungs and respiratory failure4 after thoracic surgery that may prolong the post anesthesia care unit (PACU) and hospital stays.

Although, sugammadex, a modified gamma-cyclodextrin, offers new perspectives to reduce the incidence of PORC,4 it is not available in many countries because of its significantly high cost.5

Therefore, in fast-track cardiac surgery, it seems unnecessary to maintain paralysis by repetitive bolus injection or continuous infusion of neuromuscular blockers with overall surgeons' satisfaction.6

The use of remifentanil without muscle relaxants provides excellent intubating conditions and short recovery duration.7 The effective concentration range of remifentanil for tracheal intubation without muscle relaxant is 4.5-5.5 ng/ml.8 The use of non-muscle relaxant (NMR) anesthetic techniques using remifentanil with either propofol or sevoflurane allows early extubation after trans-sternal or video-assisted thymectomy in myasthenic patients.9-10

The use of NMR technique on the surgical conditions during thoracotomy in patients without neuromuscular diseases has not yet been studied.

We hypothesizes that the use of NMR technique during thoracotomy will be associated with comparable surgical conditions with the standard use of neuromuscular blockers.

The attending anesthesiologist is not blinded. All patients will be premedicated with 1-2 mg oral lorazepam the night before surgery.

In all patients, standard monitors, and state and response entropy (SE and RE, respectively) will be applied. Neuromuscular blockade is measured with a train-of-four (TOF) (Datex-Ohmeda Division, Instrumentarium Corporation, Helsinki, Finland). The forearm is immobilized to prevent interfering movements. The ulnar nerve will be stimulated supramaximally at the wrist with a TOF stimuli (60 mA for 200 μsec) at 15-sec intervals. Baseline twitch amplitude is established after induction of anesthesia. TOF ratio is recorded as ratio between the fourth and the first twitch (T4/T1).

The radial artery is catheterized. Normothermia is maintained by using forced-air warming blankets. A thoracic epidural or paravertebral catheter is inserted but no local anesthetics are infused during the study to avoid their effects on the study outcomes.

Anesthetic technique is standardized in all studied patients. Anesthesiologists who give the anesthetic will not be involved in the collection of outcome data.

After preoxygenation, anesthesia is induced using propofol 1.5-3 mg/kg and target-controlled infusion (TCI) of remifentanil at an effect-site concentration (Ce) of 4 ng/mL using the TCI system (Injectomat® TIVA Agilia, Fresenius Kabi, France), to achieve the SE values below 50 and the difference between RE and SE below 10 and the mean arterial blood pressure (MAP) and heart rate are <20% of the baseline values. When the SE is >50 and the RE-SE difference is >10, and the MAP and heart rate are >20%, propofol 0.5 mg/kg is administered followed with gradual increases in remifentanil Ce by 0.5 ng/mL with a maximum Ce of 6 ng/ml.

Anesthesia is maintained with 0.7-1.5 minimum alveolar concentration (MAC) of sevoflurane to maintain the SE values below 50 and the difference between RE and SE below 10.

Remifentanil Ce will be increased by 0.5 ng/mL when the SE values are > 50, the difference between RE and SE >10, and the MAP and heart rate are >20% of the baseline values despite a target sevoflurane MAC ≥ 1.5.

When the SE is <50 and the RE-SE difference is <10, the sevoflurane MAC will be gradually decreased to a minimum of 0.7, followed with gradual decreases in remifentanil Ce by 0.5 ng/mL with a minimum Ce of 1.5 ng/ml.

Light anesthesia is defined as an episode with SE values that exceeds 50 and/or MAP and HR values that exceeds the baseline by 20% and that lasted for more than 3 consecutive min.

Patients' two lungs (TLV) are mechanically ventilated with fraction of inspired oxygen (FiO2) of 0.4 in air, tidal volume (VT) of 8 mL/kg, inspiratory to expiratory (I: E) ratio of 1:2.5 and PEEP of 5 cm H2O, fresh gas flow (FGF) of 1.5-1.7 l/min, and respiratory rate adjusted to achieve a PaCO2 of 35-45 mm Hg.

After pleurotomy, the patient's dependent lung is ventilated with a TV of 6 mL/kg and FiO2, I: E ratio, PEEP, FGF, and respiratory rate, are maintained as during TLV and the lumen of the nondependent lung is left open to air.

Hemodynamic control is standardized according to the authors' protocol.

During surgery, the authors will administer Lactated Ringer's solution at a rate of 2 mL/kg/h. If MAP drops down to 60 mmHg, 250 mL of plasma protein fraction 5% will be administered, and, if this is not enough, repeated doses of intravenous of ephedrine 5 mg or norepinephrine 5 µg, will be administered to maintain urine output to be equal or greater than 0.5 ml/kg/hour. A hemoglobin concentration of 8 g/dL or greater is compensated with red blood cell concentrates.

All surgical procedures will be performed by the same surgeons who are blinded for the study.

In the case of clinically unacceptable laryngoscopy and intubating conditions, poor or extremely poor surgical conditions, or a sudden deterioration of surgical conditions despite the SE values below 50, the difference between RE and SE < 10, the MAP and heart rate are <20% of the baseline values, cisatracurium is administered in a bolus dose of 0.1 mg/kg.

At the end of surgery, the nondependent lung is re-expanded, TLV is resumed as before surgery. The remifentanil and sevoflurane will be discontinued after chest closure and skin closure (T0), respectively. In the Muscle Relaxant group, during skin closure, when the TOF ratio ranged between 0.3 and 0.5, the neuromuscular blockade is antagonized with 50 µg/kg neostigmine and 10 µg/kg glycopyrrolate.

Tracheal extubation will be performed immediately when all extubation criteria were achieved (TOF ratio ≥ 0.9, spontaneous ventilation, the ability to follow verbal commands, eyes opening, head lift ≥ 5 s, and hand grip).

A pilot study showed that the proportion of the surgeons who rated their satisfaction with surgical conditions as an excellent (Score 4) in anesthetized patients with cisatracurium was 92.5%. A priori power analysis indicated that a sample size of 30 patients was sufficiently large to detect a 30% difference in the proportion of the excellent operative conditions, during the use of NMRT, a type-I error of 0.05 and a power of 90%. We added more patients (10%) for a final sample size of 33 patients to compensate patients dropping out during the study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class (II-III)
* elective open thoracotomy

Exclusion Criteria:

* New York Heart Association class> II)
* Forced vital capacity < 50% of the predicted values
* Forced expiratory volume in 1 second < 50% of the predicted values
* Hepatic diseases
* Renal diseases.
* Reactive airways.
* Neuromuscular diseases.
* Asthma
* Pregnancy
* Increased risk of regurgitation
* Anticipated difficult intubation
* Body mass index >35 kg/m2
* Electrolytes abnormalities
* Acid base abnormalities
* Repeat surgery
* history of head and neck surgery
* Preoperative circulatory support
* Preoperative ventilatory support
* Medications affecting the neuromuscular junctions
* Family history of malignant hyperthermia
* Allergy to any of the study drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Modified surgical rating scale | for 3 hours after start of surgery
  A four-point ordinal scale adopted from the surgical rating scale of Martini et al.,ranging from 1 (extremely poor conditions) to 4 (optimal conditions).
  Extremely poor (Score 1) indicates that the surgeon is unable to work because of coughing, bucking, diaphragmatic contractions or movements, or the inability to spread or approximate the ribs during chest opening and closure, respectively, because of inadequate muscle relaxation;
  poor (Score 2) indicates that there is a visible field, but the surgeon is severely hampered by continuous muscle contractions, spontaneous movements of the surgical lung, or both that could cause hazard of tissue damage;
  good (Score 3) indicates that there is an acceptable field with sporadic muscle contractions causing some interference with the surgeon's work;
  excellent (Score 4) indicates a wide working field without any lung movement or muscle contractions.

SECONDARY OUTCOMES:
heart rate | 5 min after induction of anesthesia, 1 min after chest opening, 30 min after start of surgery, 60 min after start of surgery, 90 min after start of surgery, 120 min after start of surgery, 1 min after start of chest closure, 5 min after extubation
  heart rate
Mean blood pressure | 5 min after induction of anesthesia, 1 min after chest opening, 30 min after start of surgery, 60 min after start of surgery, 90 min after start of surgery, 120 min after start of surgery, 1 min after start of chest closure, 5 min after extubation
  Mean blood pressure
Train-of-four ratio | 5 min after induction of anesthesia, 1 min after chest opening, 30 min after start of surgery, 60 min after start of surgery, 90 min after start of surgery, 120 min after start of surgery, 1 min after start of chest closure, 5 min after extubation
  Train-of-four ratio
laryngoscopy conditions | 1 min after laryngscopy
  laryngoscopy conditions
intubating conditions | 1 min after intubation
  intubating conditions
Cost of medications | after surgery
  cost of the used medications
Need for vasoactive drugs | for 3 hour during surgery
  use of ephedrine, and norepinephrine
Recovery Times | for 1 hours after surgery
  the times to spontaneous eye opening, obey verbal command, tracheal extubation and post-anesthesia care unit discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Principal Investigator — Associate Professor at Anesthesiology Dept; Mohamed A Regal, MD, Study Chair — Imam Abdulrahman Bin Faisal University
Locations (1):
- Dammam University, Khobar, Eastern Province, Saudi Arabia